CLINICAL TRIAL: NCT02492035
Title: Lifestyle Intervention for Treating Systemic Hypertension in Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Fondation IUCPQ (Other); CSSS-VC (Unknown); GMF-UMF Laval-Québec (Unknown)
Responsible Party: Principal Investigator, Caroline, MD,PhD, clinical researcher, Laval University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 20805
Record Dates: First submitted 2015-06-03; First posted 2015-07-08 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Hypertension
Keywords: Hypertension; lifestyle; clinical trials; primary care setting
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator

ARMS (4):
- Physical activity (Experimental): Tailoring intervention with kinesiologist
  Interventions: Behavioral: Lifestyle intervention
- Diet (Experimental): Tailoring intervention with nutritionist
  Interventions: Behavioral: Lifestyle intervention
- Physical activity and diet (Experimental): Tailoring intervention with kinesiologist and nutritionist
  Interventions: Behavioral: Lifestyle intervention
- Standard medical care (No Intervention): Follow with family doctor as usual care.

INTERVENTIONS:
Behavioral: Lifestyle intervention
  Arms: Diet; Physical activity; Physical activity and diet

SUMMARY:
The Canadian hypertension education program recommends increased physical activity, adoption of the Dietary Approaches to Stop Hypertension (DASH) diet, and reduction in sodium and alcohol intake for treatment and prevention of hypertension. Objective: To describe patients participating in an interdisciplinary lifestyle intervention to reduce blood pressure in a family medicine primary care setting. Design: Descriptive study. Participants: The study aims to recruit 60 sedentary hypertensive patients to participate in a 6-month randomized-controlled trial. To be eligible, patients must be ≥18 years of age, sedentary (7-day measured steps/day and self-report), hypertensive (based on 24-h ambulatory blood pressure measurements [ABPM]), non-smoker, non-diabetic and without dyslipidemia. Intervention: Patients are recruited by health care professionals of the family medicine unit and are thereafter randomized to one of four intervention groups: 1) standard medical care (control), 2) improved diet (DASH diet), 3) physical activity, or 4) both improved diet and physical activity. Patients are evaluated (pre, mid and post intervention), monitored, and educated by the interdisciplinary health care team that includes a physician, a kinesiologist, a nutritionist and a nurse, depending on the intervention group. T-tests and descriptive statistics were used to analyse data. This study will document the efficacy of a primary care lifestyle intervention program on cardiometabolic and hypertension risk factors.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Sedentary (7-day measured steps/day and self-report)
* Arterial hypertensive (based on 24-h ambulatory blood pressure measurements [ABPM])

Exclusion Criteria:

* secondary hypertension
* diabetes
* dyslipidemia
* cardiovascular diseases with complications
* smoker

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Rhéaume, MD,PhD, Principal Investigator — Laval University
Locations (1):
- GMF-UMF Laval-Québec, Québec, Canada